CLINICAL TRIAL: NCT02531828
Title: Expansion of Prospective Randomized Study Comparing the Polyurethane Films and Sugarcane Biopolymer Used as Dressings
Brief Title: Study Comparing the Polyurethane Films and Sugarcane Biopolymer Used as Dressings
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Polisa - Biopolímeros para Saúde (Industry)
Collaborators: Universidade Federal de Pernambuco (Other); Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Salvador Vilar Correia Lima, Associate Professor IV, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 23402513.9.0000.5208
Record Dates: First submitted 2014-06-12; First posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Wound; Rupture; Surgery; Cesarean Section
MeSH Terms: conditions — Wounds and Injuries; Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biopolymer Film (Experimental): Application of dressings for surgical correction.
  Interventions: Device: POLYSHAFT®
- Polyurethane Film, or the like (Active Comparator): Application of dressings for surgical correction
  Interventions: Device: Application of dressings for surgical correction.

INTERVENTIONS:
Device: Application of dressings for surgical correction. — Dressing for surgical correction
  Other Names: Polyurethane Film, or the like
  Arms: Polyurethane Film, or the like
Device: POLYSHAFT®
  Other Names: Biopolymer Film
  Arms: Biopolymer Film

SUMMARY:
The aim of this study is validate the use of biopolymer from sugar cane molasses film (POLYSHAFT®) a product developed in Experimental Station research laboratories (UFRPE) comparing to polyurethane film, or similar, used as a bandage after surgical correction of hypospadias, as well as other procedures. The main objective of the study is to prove the hypothesis the POLYSHAFT® presents similar or better outcomes in terms of biocompatibility, when compared to the polyurethane film when used as a bandage.

DETAILED DESCRIPTION:
Randomized controlled clinical trial. The target study population will comprise of the patients Unified Health System (SUS), the Outpatient Surgery and Pediatric Urology, Clinical Hospital of the Federal University of Pernambuco (UFPE), including children (from 01 years), adolescents and adults regardless of age, with lesions arising from the treatment of hypospadias, as well as other surgical injuries, according to the ethical principles outlined in Resolution 466 of the 2012 National Health Council.

Polyurethane films - Tegaderm ®

-The polyurethane films of sizes, 4.4 and 6.0 X 4.4 X 7.0 log National Agency of Sanitary Surveillance (ANVISA) / Health Ministry (MS) 10,002,070,019 manufactured by Minnesota Mining and Manufacturing Company (3M), with the following features: versatile and waterproof barrier against external contaminants, wraps to body contours promoting patient comfort.

Biopolymer film of sugarcane (POLYSHAFT ®)

-The biopolymer films of sugarcane will be provided by the research group biopolymer Sugarcane and the Experimental Station research laboratories (UFRPE). The biopolymer films have similar dimensions to the polyurethane film, which can be cut and adapted to the dimensions of the body of the patient.

All patients will be subjected to an interview being asked about previous surgery. The researcher will conduct physical and urological examination in determining the degree of hypospadias and / or other assessment procedure necessary for observation of the need (and display) the dressing with polyurethane film or biopolymer from sugar cane (POLYSHAFT®).

Patients will be randomly allocated to the groups: Biopolymer films with molasses sugar and polyurethane, using sealed, opaque, numbered envelopes containing computer-generated random distributions in 1:1 ratio in blocks of 10's envelopes will be opened in the operating room by a nurse while before starting the procedure.

All volunteers will be patients admitted to the pediatric surgery ward of the Clinical Hospital/UFPE and surgical procedures are carried out by the researchers. All patients will receive intravenous antibiotic prophylaxis at the beginning of the surgery as routine hospital clinics.

Patient recruitment and data analysis arising from the research will take place between August 2014 and August 2015, with the publication of the results expected in October 2015.

The follow-up evaluations of patients will be performed daily until removal of the bandage on the eighth postoperative day.

Variables together:

* Rate Biocompatibility: Assessment of adverse reactions such as irritation of the skin. The researcher through observation will issue a concept: how: No skin irritability, limited to the foreskin irritability and extended to other areas irritability.
* Degree of adherence: Assessed by the researcher through observation that deliver a concept as grip areas with detachment, grip without detachment or adhesion.
* Degree of annoyance: Patients or their caregivers respond to the questionnaire with the concept of "very upset," "little disturbed" or "not bothered" with the dressing.
* Grade adhesion and permanence "in situ" after being subjected to the action of water for cleaning three times a day. All observations from patient or their guardian who must be communicated to the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Age between 01 and 18 years and adults, regardless of age.

Exclusion Criteria:

* Patients with clinical complications or associated diseases that contraindication of surgical wound dressing.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The safety was assessed by adverse event reports, such as skin irritability next to the dressing area, categorized by feeling of warmth, itching, swelling, pain, and hyperemia.

SECONDARY OUTCOMES:
Efficacy of the Film of the Sugarcane Biopolymer | For time-to-event outcome measures, the time frame estimated was the 24 months.
  The efficacy was classified according to the grade of adhesiveness in the wound area (fully adhered, partially detached or without adhesiveness); the discomfort (described during the questionnaire as "very troubled", "troubled" or "not troubled" with the use of the dressing); and the transudation (this aspect was evaluated by the exudates drainage and its ability to retain wet).

CONTACTS AND LOCATIONS:
Overall Officials: Salvador VC Lima, Dr, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Martins AG, Lima SV, Araujo LA, Vilar Fde O, Cavalcante NT. A wet dressing for hypospadias surgery. Int Braz J Urol. 2013 May-Jun;39(3):408-13. doi: 10.1590/S1677-5538.IBJU.2013.03.15. PMID 23849573